CLINICAL TRIAL: NCT07170800
Title: A Multicenter, Open-label, Randomized, Active-controlled Clinical Study to Compare the Efficacy and Safety of Different Combination Regimens of JDB0131 Benzenesulfonate Tablets With Delamanid in Patients With Rifampin-resistant Tuberculosis (JD-RISE)
Brief Title: A Phase 2b Clinical Study of JDB0131 Benzenesulfonate Tablets
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: WestVac Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JDB-131-202
Record Dates: First submitted 2025-09-03; First posted 2025-09-12 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Tuberculosis; Multidrug Resistant Pulmonary Tuberculosis; Rifampicin-resistant Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — OPC-67683; Fumigant 93

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: BJLLfx(M)/C (Experimental): Bedaquiline (B) and JDB0131 (J) and Linezolid (L) and Levofloxacin (Lfx) or (Moxifloxacin (M)) / Clofazimine (C)
  Patients will take medications for 8 consecutive weeks.
  Patients will be randomized based on fluoroquinolone resistance. If fluoroquinolone-susceptible, patients in group A will receive Levofloxacin (Lfx) or Moxifloxacin (M). If fluoroquinolone-resistant, patients in group A will receive Clofazimine （C）.
  Interventions: Drug: JDB0131 100mg
- Group B: BJLLfx(M)/C (Experimental): Bedaquiline (B) and JDB0131 (J) and Linezolid (L) and Levofloxacin (Lfx) or (Moxifloxacin (M)) / Clofazimine (C).
  Patients will take medications for 8 consecutive weeks.
  Patients will be randomized based on fluoroquinolone resistance. If fluoroquinolone-susceptible, patients in group A will receive Levofloxacin (Lfx) or Moxifloxacin (M). If fluoroquinolone-resistant, patients in group A will receive Clofazimine （C）.
  Interventions: Drug: JDB0131 200mg
- Group C: BDLLfx/C (Active Comparator): Bedaquiline (B) and Delamanid (D) and Linezolid (L) and Levofloxacin (Lfx) / Clofazimine (C).
  Patients will take medications for 8 consecutive weeks.
  Patients will be randomized based on fluoroquinolone resistance. If fluoroquinolone-susceptible, patients in group C will receive Levofloxacin (Lfx). If fluoroquinolone-resistant, patients in group C will receive Clofazimine (C).
  Interventions: Drug: Delamanid (D)

INTERVENTIONS:
Drug: JDB0131 100mg — Bedaquiline (B): For the first 2 weeks, 400 mg qd; then adjust to 200 mg tiw.
  JDB0131 (J): 100 mg bid.
  Linezolid (L): 600 mg qd.
  Levofloxacin (Lfx): According to body weight, patients ≤50 kg, 750 mg qd; patients >50 kg, 1000 mg qd.
  Moxifloxacin (M): 400 mg qd.
  Clofazimine (C): 100 mg qd.
  Arms: Group A: BJLLfx(M)/C
Drug: JDB0131 200mg — Bedaquiline (B): For the first 2 weeks, 400 mg qd; then adjust to 200 mg tiw.
  JDB0131 (J): 200 mg bid.
  Linezolid (L): 600 mg qd.
  Levofloxacin (Lfx): According to body weight, patients ≤50 kg, 750 mg qd; patients >50 kg, 1000 mg qd.
  Moxifloxacin (M): 400 mg qd.
  Clofazimine (C): 100 mg qd.
  Arms: Group B: BJLLfx(M)/C
Drug: Delamanid (D) — Bedaquiline (B): For the first 2 weeks, 400 mg qd; then adjust to 200 mg tiw.
  Delamanid (D): 100 mg bid.
  Linezolid (L): 600 mg qd.
  Levofloxacin (Lfx): According to body weight, patients ≤50 kg, 750 mg qd; patients >50 kg, 1000 mg qd.
  Moxifloxacin (M): 400 mg qd.
  Clofazimine (C): 100 mg qd.
  Arms: Group C: BDLLfx/C

SUMMARY:
This is a multicenter, randomized, open-label, active-controlled clinical study designed to evaluate the efficacy, safety, and pharmacokinetic characteristics of different doses of JDB0131 benzenesulfonate tablets compared with delamanid in combination with bedaquiline, linezolid, levofloxacin (moxifloxacin)/clofazimine, etc. in the treatment of patients with drug-resistant (including rifampicin-resistant) tuberculosis for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age: 14 years through 65 years of age, male or female
* Weight: 40kg ≤ weight ≤ 90kg
* Patients with clinically confirmed pulmonary tuberculosis, Drug Susceptibility Testing (DST) results confirmed to be at least rifampicin-resistant, molecular or phenotypic DST results within 3 months before enrollment can be received
* Sputum acid-fast bacilli smear is positive (≥2+ once or 1+ twice at least)
* Patients who are currently taking anti-tuberculosis treatment or using drugs with anti-tuberculosis effects agree to stop all anti-tuberculosis drug treatment and complete a 7-day washout period
* Women of reproductive age must agree to use highly effective contraceptive measures throughout the study and for at least 6 months after discontinuation of the drug. Male participants whose partners are women of reproductive age must agree to use appropriate contraceptive methods throughout the study and for at least 6 months after discontinuation of the drug (see protocol Appendix 1)
* Fully understand the purpose and requirements of this trial, voluntarily sign the written informed consent and agree to abide by the relevant provisions of the informed consent

Exclusion Criteria:

* Those who cannot take delamanid, bedaquiline, or linezolid for various reasons
* Take delamanid, bedaquiline, or linezolid for more than 1 month (can be enrolled if evidence of no resistance to the above drugs is provided)
* Hematogenously disseminated pulmonary tuberculosis or severe extrapulmonary tuberculosis as determined by the investigator; or patients with pulmonary tuberculosis who are assessed by the investigator to be likely to require surgical treatment within 8 weeks
* History of torsades de pointes or risk factors, including a personal or family history of long QT syndrome (LQTS), persistent hypothyroidism, or bradycardia
* Anyone with any of the following cardiovascular diseases or other conditions within 6 months before enrollment:

  1. Myocardial infarction;
  2. Heart surgery or coronary revascularization (coronary artery bypass grafting/percutaneous transluminal coronary angioplasty);
  3. Unstable angina;
  4. Congestive heart failure (New York Heart Association functional class III or IV);
  5. Transient ischemic attack or severe cerebrovascular disease.
* Peripheral neuropathy CTCAE grade 3 or 4; Grade 1 or 2 peripheral neuropathy that the investigator judges may progress/worsen during the study; Patients with optic neuritis
* History of gastrointestinal surgery or resection that may affect the absorption and/or excretion of oral medications
* Patients who are considered by the investigator to be unsuitable for this trial due to unstable or severe cardiovascular, renal, hepatic, blood, tumor, endocrine metabolic, psychiatric or rheumatic diseases
* History of alcohol dependence or drug abuse within 6 months before screening, the investigator believes that it may affect the safety of the participants and affect the trial compliance
* Patients who have used other clinical trial investigational drugs within 3 months before administration
* Concomitant take drugs that cause bone marrow suppression
* Concomitant take serotonin reuptake inhibitors, tricyclic antidepressants, serotonin, serotonin receptor agonists, and other drugs
* Concomitant take drugs that prolong the QT interval, such as quinidine, procainamide, amiodarone, sotalol, etc.
* Chronic systemic corticosteroid therapy, cumulative take for more than 4 weeks within 3 months before enrollment
* Allergic to any investigational drug or related substance as confirmed by the researcher's clinical judgment
* Women who have a positive pregnancy test during screening or are breastfeeding
* Patients with hepatitis B virus (HBV) positive results (HBsAg, HBeAg, and HBcAb); positive hepatitis C virus (HCV) antibodies and aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels >3 times the upper limit of normal; positive Human Immunodeficiency Virus (HIV) antibody test; positive syphilis antibody test and active syphilis
* Laboratory tests show any of the following:

  1. Hemoglobin < 80 g/L;
  2. platelets < 75 ✕ 109 /L;
  3. Aspartate aminotransferase (AST) > 3 times the upper limit of normal;
  4. Alanine aminotransferase (ALT) > 3 times the upper limit of normal;
  5. Serum total bilirubin (TBIL) > 2 times the upper limit of normal;
  6. Serum creatinine (Cr) > 1.5 times the upper limit of normal;
  7. Serum amylase > 2 times the upper limit of normal.
* The following abnormalities were found in the electrocardiogram (ECG):

  1. At least twice QTcF intervals > 450 ms (male) or > 470 ms (female);
  2. Pathological Q waves (defined as >40 ms or deep >0.4-0.5mV);
  3. ECG suggests preexcitation syndrome;
  4. ECG suggests left bundle branch block or right bundle branch block; or second or third degree heart block;
  5. Intraventricular conduction delay with QRS duration >120ms;
  6. Bradycardia with a sinus rate < 50 bpm.
* In the investigator's judgment, any condition that affects the subject's compliance with the study protocol, or any serious medical or psychological condition that may affect the interpretation of efficacy and safety data, or any condition that may affect the subject's safety when participating in the trial

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-09-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients with Sputum Culture Conversion (SCC) | During the 8-week treatment period and after treatment
  SCC was defined as a patient without SCC at baseline who subsequently met the definition of SCC. A patient was classified as having achieved SCC if he/she achieved 2 consecutive sputum cultures negative for growth of mycobacterium tuberculosis (MTB) at least 7 days apart and had no further sputum cultures that were positive for growth within the specified time frame. Patients who have sputum cultures that were positive during treatment but only converted to negative at the end of treatment were also counted as negative.

SECONDARY OUTCOMES:
Time to Sputum Culture Conversion (SCC) | During the 8-week treatment period and after treatment
  SCC was defined as a patient without SCC at baseline who subsequently met the definition of SCC. A patient was classified as having achieved SCC if he/she achieved 2 consecutive sputum cultures negative for growth of mycobacterium tuberculosis (MTB) at least 7 days apart and had no further sputum cultures that were positive for growth within the specified time frame. Patients who have sputum cultures that were positive during treatment but only converted to negative at the end of treatment were also counted as negative.
  Time to SCC was defined as the earliest time of two consecutive sputum cultures negative for growth, that is, the time (specimen collection time) of the first sputum culture negative for growth among two consecutive sputum cultures negative for growth of mycobacterium tuberculosis (MTB) at least 7 days apart was taken as the negative conversion time, expressed in days.
Time to positivity (TTP) | During the 8-week treatment period and after treatment
  Time-to-positivity (TTP) is defined as the length of time from the beginning of culture incubation to the positive detection of mycobacterium tuberculosis growth.
Number of Participants With Clinically Significant Abnormality in Vital Signs | During the 8-week treatment period
  Vital signs included body temperature (degree Celsius), heart rate [beats/minute (bpm)], breathe [times/minute (tpm)], systolic and diastolic blood pressure [millimetre of mercury (mm Hg)].
Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG) Values | During the 8-week treatment period
  The clinically significant abnormal ECG values including ventricular rate outlier, PR outlier, QRS outlier, QT outlier and QTcF outlier.
Number of Participants With Clinical Significant Abnormality in Laboratory Test | During the 8-week treatment period
  Laboratory assessments included parameters for serum chemistry (Aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, lactate dehydrogenase, glutamyl transpeptidase, total bilirubin, direct bilirubin, sodium, potassium, chlorine, urea, creatinine), hematology (Red blood cell count, hemoglobin concentration, mean corpuscular volume, white blood cell count, platelet count, neutrophil count, lymphocyte count, monocyte count, eosinophil count, basophil count), urinalysis (Urine leukocytes, urine red blood cells, urine pH, urine specific gravity, urine protein, urine glucose, urine occult blood), stool routine (stool characteristics, stool color, fecal white blood cells, fecal red blood cells, fecal occult blood test) and other serum chemistry (specified in protocol).
Number of Patients With Adverse Events (AEs) and at least one Treatment-emergent Adverse Events (TEAEs) | During the 8-week treatment period
  An adverse event (AE) is any untoward medical occurrence in a participant/clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with treatment. A TEAE is any new AE or worsening of an existing condition after initiation of study drug.
Number of Patients With Serious Adverse Events (SAEs) | During the 8-week treatment period
  An SAE is an AE that resulted in death, inpatient hospitalization/prolongation of existing hospitalization, persistent or significant disability or incapacity, life-threatening, a congenital anomaly/birth defect, or an important medical event.
Number of Participants With Any Concomitant Medication Usage | During the 8-week treatment period
  Concomitant medications are defined as medications that started on or after the first day of study treatment or were started prior to study treatment but were ongoing on the first day of study treatment.
Time to peak (Tmax) | During the 8-week treatment period (specified in protocol)
Peak concentration (Cmax) | During the 8-week treatment period (specified in protocol)
Area under the plasma concentration-time curve from the first medication to 12 hours (AUC0-12) | During the 8-week treatment period (specified in protocol)
Time to peak at steady state (Tss,max) | During the 8-week treatment period (specified in protocol)
Peak concentration at steady state (Css,max) | During the 8-week treatment period (specified in protocol)
Trough concentration at steady state (Css,min) | During the 8-week treatment period (specified in protocol)
Average steady-state plasma concentration (Css,avg) | During the 8-week treatment period (specified in protocol)
Elimination half-life (t1/2,ss) | During the 8-week treatment period (specified in protocol)
Area under the plasma concentration-time curve from the last dose to 12 hours (AUC0-12,ss) | During the 8-week treatment period (specified in protocol)
Area under the plasma concentration-time curve from the last dose to the last measurable concentration time t (AUC0-t,ss) | During the 8-week treatment period (specified in protocol)
Area under the plasma concentration-time curve from the last dose extrapolated to infinity (AUC0-∞,ss) | During the 8-week treatment period (specified in protocol)
Apparent volume of distribution (Vd,ss/F) | During the 8-week treatment period (specified in protocol)
Oral clearance (CLss/F) | During the 8-week treatment period (specified in protocol)
Accumulation ratio: Rac(Cmax) = Cmax,ss on day 56 / Cmax on day 1 | During the 8-week treatment period (specified in protocol)
Rac (AUC) = AUC0-12,ss on day 56 / AUC0-12 on day 1 | During the 8-week treatment period (specified in protocol)
Fluctuation coefficient: fluctuation percentage at steady state = 100 * (Css,max - Css,min) / Css,avg | During the 8-week treatment period (specified in protocol)

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Wuhan Pulmonary Hospital, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - Shandong Public Health Clinical Center, Jinan, Shandong
  - Public Health Clinical Center of Chengdu, Chengdu, Sichuan
  - Beijing Chest Hospital, Capital Medical University, Beijing
  - Huashan Hospital Fudan University, Shanghai